CLINICAL TRIAL: NCT01971073
Title: Transcranial Direct Current Stimulation Influences on Cognitive Inhibition in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in financing the research
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Nira Mashal, Dr. Mashal, PI, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BARILAN-13-0116-MV-CTIL
Record Dates: First submitted 2013-10-12; First posted 2013-10-29 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia
Keywords: schizophrenic patients; tDCS; Executive functions; Dorsolateral prefrontal cortex
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bilateral Anodal-L/R Cathodal-R/L tDCS (Experimental): bilateral Anodal-left and cathodal-right tDCS over DLPFC or bilateral Anodal-right and cathodal-left tDCS over DLPFC.
  Intervention: Device: transcranial direct current stimulation
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham tDCS
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: transcranial direct current stimulation — arm Participants will receive bilateral anodal-left cathodal-right tDCS or anodal-right cathodal-left tDCS over the DLPFC.
  The following parameters will be used: stimulation intensity of 2 milliAmps for 20 minutes (6 consecutive sessions ).
  Other Names: Active Comparator: sham tDCS
  Arms: bilateral Anodal-L/R Cathodal-R/L tDCS
Device: sham tDCS — the sham tDCS group. Neuropsychological testing and symptom ratings will be conducted at baseline and 4 weeks after the end of treatment
  Arms: Sham tDCS

SUMMARY:
A deficit in cognitive suppression is a trait of patients with schizophrenia. Cognitive suppression is the ability to control or suppress irrelevant responses and to adopt relevant responses instead. The purpose of this study is to investigate the effects of transcranial direct current stimulation (tDCS) on information suppression in schizophrenic patients. This is a noninvasive technique of brain stimulation that induces prolonged functional changes in the cerebral cortex through the application of a weak direct current to the scalp (Nitsche & Paulus, 2001). The aim of this study is to test whether bilateral tDCS over the dorsolateral prefrontal cortex (DLPFC) differentially modify performance on several cognitive tasks.

DETAILED DESCRIPTION:
A deficit in cognitive suppression is a trait of patients with schizophrenia. Cognitive suppression is the ability to control or suppress irrelevant information and to adopt relevant responses instead. This ability is a basic skill which is essential to maintain a normal well-adjusted life. We need to suppress distracting information in order to focus attention, to suppress irrelevant cues in order to retrieve particular memories, and to suppress habitual responses in order to make adaptive choices (Dillon & Pizzagalli, 2007). The purpose of this study is to investigate the effects of transcranial direct current stimulation (tDCS) on information suppression in schizophrenic patients. This is a noninvasive technique of brain stimulation that induces prolonged functional changes in the cerebral cortex through the application of a weak direct current to the scalp (Nitsche & Paulus, 2001; Nitsche et al., 2003, 2004; Antal et al., 2004). The aim of this study is to test whether anodal and cathodal tDCS differentially modify performance on several cognitive tasks when applied to the left/right dorsolateral prefrontal cortex (DLPFC).

Sixty patients will be divided into four groups: 1) 15 schizophrenic subjects in a tDCS treatment group; 2) 15 schizophrenic subjects in a sham tDCS group; 3) 15 healthy subjects in a tDCS treatment group; 4) 15 healthy subjects in a sham tDCS group. All participants will complete baseline tests including an n-back test, the Hayling test and metaphoric comprehension test. The schizophrenic subjects only, will complete a bank of cognitive tests as a baseline (MATRICS Consensus Cognitive Battery (MCCB). The first meeting for the schizophrenic subjects only will be used to determine the best stimulation area (right/left DLPFC) and type (anodal/ cathodal). Schizophrenic subjects in both the treatment and the control groups will undergo six treatment sessions in total. The cognitive tests will be given to all participants once again at the end of the study. In order to evaluate improvement between the pre-test and the post-test, differences in reaction times and error rate will be calculated for each participant.

This study is important for few reasons. First, this study focus on the difficulty of suppressing irrelevant information, executive function ability essential to leading a normal life. Special populations, and specifically people with schizophrenia, have difficulty suppressing irrelevant information, and a correlation has been noted between this characteristic and weak executive functioning capabilities. In this study we evaluate the potential of minimizing these difficulties through use of tDCS. This particular tool was chosen for the study because it is easy to use, non-invasive, and painless. Research has shown that tDCS stimulation of the DLPFC can improve performance in cognitive tasks, a result that has not been mirrored through use of medications. Second, in recognition of the heterogeneity of schizophrenic patients (substantiated by the fact that the success of other treatments varies from patient to patient), our study will perform tests to identify the preferred stimulation region, DLPFC left/right. The results will help determine more specifically if there is a degree of heterogeneity in terms of the region responsible for suppressing irrelevant information . Related to this, we will be able to assess the impact of stimulation, including whether or not stimulation benefits all schizophrenic patients or, alternatively, if there are unknown variables involved which determine the relative success of this treatment amongst individuals. In addition, we will be able to explore differences or correlations between healthy subjects' verbal abilities in relation to the various tests conducted, and assess the impact of these tests on healthy subjects' cognitive inhibition and working memory. Finally, this study is critical because if the treatment method proves to be successful, we would be able to extend this study to other populations that have difficulties with executive functioning, and in addition, to examine the effect of electrical stimulation on other cognitive abilities.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years old or above.
* Clinical diagnosis of schizophrenia or schizoaffective disorder
* must be with a stable mental status as demonstrated by a stable Positive and -Negative Symptom Score (PANSS) score over a period of 2 weeks.
* must have no medication changes in the 2 weeks prior to obtaining informed consent.
* must be able to give informed consent for the trial.

Exclusion Criteria:

* Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
* Pregnant or breast-feeding.
* current DSM-V substance or alcohol abuse.
* Concurrent delirium
* mental retardation
* drug-induced psychosis
* history of clinically significant brain trauma documented by CT or MRI.
* epilepsy or had seizures 6 months prior the beginning of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Progression score on cognitive tasks | two years
  Improve performance in cognitive tasks in particular, higher scores on the MATRICS Consensus Cognitive Battery in the post vs. before intervention tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nira Mashal, Ph.D., Principal Investigator — Bar Ilan University
Locations (1):
- The Chaim Sheba Medical Center, Ramat Gan, Israel